CLINICAL TRIAL: NCT07112157
Title: Efficacy of Oxalidine and Sufentanil in Strabismus Correction: a Non Inferiority Trial
Brief Title: Efficacy of Oxalidine and Sufentanil in Strabismus Correction
Acronym: strabismus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HenanPPH-FNN3
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Strabismus Surgery
Keywords: strabismus surgery; analgesia
MeSH Terms: conditions — Agnosia | interventions — ((3-methoxythiophen-2-yl)methyl)((2-(9-(pyridin-2-yl)-6-oxaspiro(4.5)decan-9-yl)ethyl))amine; Sufentanil

STUDY DESIGN:
Intervention Model Description: The purpose of this trial is to compare the analgesic effect of oxalidine and sufentanil in strabismus surgery, verify that the analgesic effect of oxalidine is not inferior to sufentanil, and evaluate the safety of the two drugs and the impact on postoperative recovery.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oliceridine group (Experimental): After entering the room, the patient was intravenously injected with oselidine at a dose of 0.08mg/kg during anesthesia induction
  Interventions: Drug: Oliceridine
- Sufentanil group (Active Comparator): After the patient entered the room, sufentanil was injected intravenously during anesthesia induction with a dose of 0.4 μ g/kg
  Interventions: Drug: Sulfentanil

INTERVENTIONS:
Drug: Oliceridine — After entering the room, the patient was intravenously injected with oselidine at a dose of 0.08mg/kg during anesthesia induction
  Arms: Oliceridine group
Drug: Sulfentanil — After the patient entered the room, sufentanil was injected intravenously during anesthesia induction with a dose of 0.4 μ g/kg
  Arms: Sufentanil group

SUMMARY:
The purpose of this study is to compare the anesthetic effect of oxalidine and sufentanil in strabismus surgery through a non inferiority test, including analgesic efficacy, intraoperative hemodynamic stability, postoperative recovery quality and the incidence of adverse reactions. . This study will provide a new evidence-based basis for the application of opioids in ophthalmic short surgery, and may improve the perioperative experience of patients.

DETAILED DESCRIPTION:
Since surgery involves fine manipulation of the ocular muscles, postoperative pain and oculocardiac reflex (OCR) are common clinical challenges. Therefore, anesthesia management should not only ensure adequate analgesia, but also minimize stress reactions and adverse reactions caused by surgical stimuli. At present, opioids such as sufentanil are widely used in the anesthesia scheme of such surgery because of its potent analgesia and stable hemodynamic characteristics. However, sufentanil may cause respiratory depression, postoperative nausea and vomiting (PONV) and other side effects, and its high lipid solubility may prolong the postoperative recovery time.

Oliceridine is a new selective μ - opioid receptor agonist. Compared with traditional opioids, it has the characteristics of biased activation of G protein pathway, which may provide effective analgesia and reduce the adverse reactions mediated by β - arrestin pathway (such as respiratory depression and gastrointestinal dysfunction). Recent studies have shown that oselidine has shown good safety and efficacy in postoperative analgesia, but its application in short ophthalmic surgery (such as strabismus correction) has not been fully explored.

ELIGIBILITY:
Inclusion Criteria:

* The patients to be treated with strabismus correction under general anesthesia are 3-60 years old, regardless of gender.

The American Society of anesthesiologists (ASA) classification is Ⅰ - Ⅱ. Patients or their guardians (for child patients) voluntarily participated in the trial and signed the informed consent form with informed consent.

Exclusion Criteria:

* Those who are allergic to oxalidine, sufentanil or any of the ingredients in their preparations.

Patients with severe heart, liver, kidney and other important organ dysfunction.

Have a history of epilepsy or central nervous system disease. Other opioid analgesics were used within 48 hours before operation. Pregnant or lactating women. Patients with mental disorders who are unable to cooperate to complete the test related assessment.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 290 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adequate rate of intraoperative analgesia | From enrollment to the end of treatment at 1 day
  Definition: No body movement (body movement score ≤ 1) and no need for additional analgesics during surgical skin cutting and eye muscle traction.
  Evaluation method:
  Physical activity score (0-3 points): 0=none; 1=Mild (does not interfere with surgery); 2=Obvious (requiring intervention); 3=Severe (pause surgery).
Success rate of initial insertion of laryngeal mask | From enrollment to the end of treatment at 1 day
  One time insertion of laryngeal mask without adjustment/replacement, and good airway sealing (normal ETCO ₂ waveform)

SECONDARY OUTCOMES:
Ocular Heart Reflex (OCR) incidence rate | From enrollment to the end of treatment at 1 day
  HR decline>20% may require atropine intervention.
Hemodynamic fluctuations | From enrollment to the end of treatment at 1 day
  Hypotension (MAP<65 mmHg or decrease from baseline>30%), hypertension (MAP>100 mmHg)
Respiratory inhibition: | From enrollment to the end of treatment at 1 day
  SpO ₂<90% or ETCO ₂>50 mmHg
Postoperative nausea and vomiting (PONV) (0-24h) | From enrollment to the end of treatment at 1 day
  Rating: 0=none; 1=Mild (no need for treatment); 2=Moderate (requires antiemetic medication); 3=Severe (repeated vomiting)

IPD SHARING:
Plan to Share IPD: No